CLINICAL TRIAL: NCT03321214
Title: A Pilot Study to Test the Feasibility and Acceptability of Using a Gluten Sensor Device to Promote Gluten Free Diet Adherence and Quality of Life in Patients With Celiac Disease
Brief Title: Gluten Sensor Device to Promote Gluten Free Diet Adherence and Quality of Life in Patients With Celiac Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAR6004
Record Dates: First submitted 2017-10-20; First posted 2017-10-25 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Celiac Disease
Keywords: Gluten Free diet
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Light use of Nima (Experimental): Ten participants will be randomized to receive 12 capsules every other month (18 capsules for the 3 months which is considered light use).
  Interventions: Other: Gluten Sensor Dose-Finding Intervention
- Moderate use of Nima (Experimental): Ten participants will be randomized to receive 12 capsules per month (36 capsules for the 3 months which is considered moderate use).
  Interventions: Other: Gluten Sensor Dose-Finding Intervention
- Heavy use of Nima (Experimental): Ten participants will be randomized to receive 24 capsules per month (72 capsules for the 3 months which is considered heavy use).
  Interventions: Other: Gluten Sensor Dose-Finding Intervention

INTERVENTIONS:
Other: Gluten Sensor Dose-Finding Intervention — Nima is a small portable sensor that detects gluten in a small amount of liquid and solid foods in about three minutes. Nima combines an electronic sensor with antibody-based detection in a disposable capsule. Nima displays a "smiley face" if the food or beverage is < 20 ppm or a wheat icon for > 20 ppm (low or high gluten).
  Each of the 30 participants will receive a Nima along with 3 months of disposable capsules. At the baseline visit, research staff will provide participants with the Nima and capsules and review instructions on how to properly use the device with all participants.
  Other Names: Nima

SUMMARY:
The current treatment for celiac disease is a strict 100% gluten free diet. Little is known about the best way to promote adherence to such a strict diet and how to maximize quality of life at the same time.

This pilot will look at the utility of a new innovation to promote gluten free diet adherence - a portable gluten sensor device. Participants will be 30 teenagers and adults with celiac disease recruited from the Celiac Disease Center at Columbia University in New York City. Before and after the intervention, participants will be asked about their adherence to a gluten free diet, quality of life, symptoms, and feelings of anxiety, and depression. This pilot data will help to inform interventions that the investigators hope to test in a larger NIH-funded trial to better understand the best ways to promote adherence and quality of life in celiac patients.

DETAILED DESCRIPTION:
Little is known about the best ways to promote a strict gluten-free diet while maximizing quality of life in teenagers and adults with celiac disease. The aim of the proposed pilot is to assess the acceptability and feasibility of a novel intervention - a portable gluten sensor device. The sample for this pilot will be 30 teenagers and adults with biopsy confirmed celiac disease recruited from the Celiac Center at Columbia University in New York City. Thirty participants will pilot test a portable gluten sensor device with its associated iPhone app for 3 months. At baseline and three-month follow-up, participants will complete measures of gluten free diet adherence, quality of life,symptoms, anxiety, and depression. At post-only, the investigators will collect in-depth data related to the feasibility and acceptability of the gluten sensor, as well as facilitators and barriers related to how, where, and when it was used. At the completion of the proposed pilot study, the investigators hope to have preliminary data to inform development of gluten sensor interventions that the investigators hope to test in a larger NIH-funded randomized controlled trial. These findings, in combination with a larger trial, have the potential for the development of a new standard of care in the management of patients with celiac disease.

ELIGIBILITY:
Inclusion Criteria:

* Individuals >13 years old (15 teenagers and 15 adults), 30 in total with duodenal biopsy-confirmed diagnosis of celiac disease will be recruited to participate.
* As we are testing a gluten sensor device, we require that participants are 13 years or older as they will need to be able to operate the gluten sensor device independently

Exclusion Criteria:

* No participants will be excluded based on gender, race or ethnicity.
* Patients diagnosed with celiac disease without a duodenal biopsy.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Quality of life measure | 3 months
  A 20-item Celiac Disease-Quality of Life (CD-QOL) survey or 17-item Celiac Disease Pediatric Quality of (CDPQOL) survey. Each of these scales ranges from a minimum of 0 (lowest quality of life) to 100 (highest quality of life).

SECONDARY OUTCOMES:
Depression | 3 months
  The 21 item Beck Depression Inventory (BDI). This depression scale ranges from 0 (fewer symptoms) to 60 (most symptoms).
Adherence to the gluten-free diet | 3 months
  A 7-item validated CD adherence test (CDAT) survey. Higher scores suggest worse adherence (with scores >13 indicative of poor adherence)
Celiac disease symptoms | 3 months
  Celiac Disease Symptom Diary (CDSD)
Anxiety | 3 months
  21 item Beck Anxiety Inventory. This anxiety index ranges from 20 (lower anxiety) to 100 (greater anxiety).

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Lebwohl, MD,MS, Principal Investigator — Columbia University
Locations (1):
- Celiac Disease Center at Columbia University, New York, New York, United States

REFERENCES:
- [Background] Green PHR, Krishnareddy S, Lebwohl B. Clinical manifestations of celiac disease. Dig Dis. 2015;33(2):137-140. doi: 10.1159/000370204. Epub 2015 Apr 22. PMID 25925914
- [Background] Abu Daya H, Lebwohl B, Lewis SK, Green PH. Celiac disease patients presenting with anemia have more severe disease than those presenting with diarrhea. Clin Gastroenterol Hepatol. 2013 Nov;11(11):1472-7. doi: 10.1016/j.cgh.2013.05.030. Epub 2013 Jun 10. PMID 23756221
- [Background] Rubio-Tapia A, Kyle RA, Kaplan EL, Johnson DR, Page W, Erdtmann F, Brantner TL, Kim WR, Phelps TK, Lahr BD, Zinsmeister AR, Melton LJ 3rd, Murray JA. Increased prevalence and mortality in undiagnosed celiac disease. Gastroenterology. 2009 Jul;137(1):88-93. doi: 10.1053/j.gastro.2009.03.059. Epub 2009 Apr 10. PMID 19362553
- [Background] Rubio-Tapia A, Ludvigsson JF, Brantner TL, Murray JA, Everhart JE. The prevalence of celiac disease in the United States. Am J Gastroenterol. 2012 Oct;107(10):1538-44; quiz 1537, 1545. doi: 10.1038/ajg.2012.219. Epub 2012 Jul 31. PMID 22850429
- [Background] Lohi S, Mustalahti K, Kaukinen K, Laurila K, Collin P, Rissanen H, Lohi O, Bravi E, Gasparin M, Reunanen A, Maki M. Increasing prevalence of coeliac disease over time. Aliment Pharmacol Ther. 2007 Nov 1;26(9):1217-25. doi: 10.1111/j.1365-2036.2007.03502.x. PMID 17944736
- [Background] Meyer D, Stavropolous S, Diamond B, Shane E, Green PH. Osteoporosis in a north american adult population with celiac disease. Am J Gastroenterol. 2001 Jan;96(1):112-9. doi: 10.1111/j.1572-0241.2001.03507.x. PMID 11197239
- [Background] Lebwohl B, Granath F, Ekbom A, Smedby KE, Murray JA, Neugut AI, Green PH, Ludvigsson JF. Mucosal healing and risk for lymphoproliferative malignancy in celiac disease: a population-based cohort study. Ann Intern Med. 2013 Aug 6;159(3):169-75. doi: 10.7326/0003-4819-159-3-201308060-00006. PMID 23922062
- [Background] Hall NJ, Rubin G, Charnock A. Systematic review: adherence to a gluten-free diet in adult patients with coeliac disease. Aliment Pharmacol Ther. 2009 Aug 15;30(4):315-30. doi: 10.1111/j.1365-2036.2009.04053.x. Epub 2009 May 26. PMID 19485977
- [Background] Comino I, Fernandez-Banares F, Esteve M, Ortigosa L, Castillejo G, Fambuena B, Ribes-Koninckx C, Sierra C, Rodriguez-Herrera A, Salazar JC, Caunedo A, Marugan-Miguelsanz JM, Garrote JA, Vivas S, Lo Iacono O, Nunez A, Vaquero L, Vegas AM, Crespo L, Fernandez-Salazar L, Arranz E, Jimenez-Garcia VA, Antonio Montes-Cano M, Espin B, Galera A, Valverde J, Giron FJ, Bolonio M, Millan A, Cerezo FM, Guajardo C, Alberto JR, Rosinach M, Segura V, Leon F, Marinich J, Munoz-Suano A, Romero-Gomez M, Cebolla A, Sousa C. Fecal Gluten Peptides Reveal Limitations of Serological Tests and Food Questionnaires for Monitoring Gluten-Free Diet in Celiac Disease Patients. Am J Gastroenterol. 2016 Oct;111(10):1456-1465. doi: 10.1038/ajg.2016.439. Epub 2016 Sep 20. PMID 27644734
- [Background] Silvester JA, Graff LA, Rigaux L, Walker JR, Duerksen DR. Symptomatic suspected gluten exposure is common among patients with coeliac disease on a gluten-free diet. Aliment Pharmacol Ther. 2016 Sep;44(6):612-9. doi: 10.1111/apt.13725. Epub 2016 Jul 22. PMID 27443825
- [Derived] Wolf RL, Vipperman-Cohen A, Green PHR, Lee AR, Reilly NR, Zybert P, Lebwohl B. Portable gluten sensors: qualitative assessments by adults and adolescents with coeliac disease. J Hum Nutr Diet. 2020 Dec;33(6):876-880. doi: 10.1111/jhn.12810. Epub 2020 Sep 25. PMID 32975829
- [Derived] Wolf RL, Green PHR, Lee AR, Reilly NR, Zybert P, Lebwohl B. Benefits From and Barriers to Portable Detection of Gluten, Based on a Randomized Pilot Trial of Patients With Celiac Disease. Clin Gastroenterol Hepatol. 2019 Nov;17(12):2605-2607. doi: 10.1016/j.cgh.2019.03.011. Epub 2019 Mar 15. PMID 30885882